CLINICAL TRIAL: NCT04562649
Title: Community Health Worker And MHealth to ImProve Viral Suppression
Acronym: CHAMPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Rebecca Schnall, RN, MPH, PhD, Mary Dickey Lindsay Professor of Disease Prevention and Health Promotion, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AAAT2430; R01NR019758 (NIH)
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: HIV/AIDS
Keywords: ART; PLWH
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention (Experimental): Wise App that delivers medication adherence reminders and community health worker sessions
  Interventions: Device: Wise App with medication adherence reminders; Behavioral: CHW Sessions
- Control (No Intervention): Standard of care

INTERVENTIONS:
Device: Wise App with medication adherence reminders — The Intervention group will receive the Wise App that delivers medication adherence reminders.
  Arms: Intervention
Behavioral: CHW Sessions — The Intervention group will complete sessions with a community health worker (CHW).
  Arms: Intervention

SUMMARY:
The overall goal of this study is to evaluate the effects of the CHAMPS intervention for people living with HIV (PLWH) in a randomized controlled trial. The proposed trial is scientifically significant in representing a principled and systematic effort to test the efficacy of a combined community health worker (CHW) and smartphone intervention linked to a smart pill box for antiretroviral (ART) adherence in PLWH in the United States (US). Guided by a rigorous theoretical model of supportive accountability and building on preliminary work, this intervention has the potential to enable PLWH to self-manage their ART regimens while CHW monitor their ART adherence in real-time ultimately leading to viral suppression and ART adherence.

DETAILED DESCRIPTION:
Persons living with HIV (PLWH) now achieve a near-normal life expectancy due to antiretroviral therapy (ART) which has transformed HIV from a terminal diagnosis to a manageable chronic condition. Despite widespread availability of ART in the United States (US), many of the country's approximate 1.1 million PLWH are not fully benefitting from ART due to poor adherence. These suboptimal HIV health outcomes occur at a time when clinicians have limited time and the US healthcare system remains fragmented, further exacerbating the challenges inherent in the lives of underserved, marginalized groups, such as PLWH. Therefore, the development and evaluation of interventions using a cadre of community health workers (CHW) holds promise for addressing these challenges in the US. This study addresses limitations in current research on CHW interventions to improve viral suppression and ART adherence. The investigators propose to build on strong preliminary data to strengthen a community health worker (CHW) intervention using an existing mHealth approach, and provide further information regarding the successful wide-scale implementation of this combination intervention.

ELIGIBILITY:
Inclusion Criteria:

* Be able to communicate and read in English or Spanish
* Willing to participate in any assigned arm of the intervention
* Diagnosed with HIV ≥6 months ago
* Have an HIV-1 RNA level >200 copies/mL, or have at least one "no-show" visit in the past 12 months, or report being virally unsuppressed in the past 12 months
* Have ART adherence <80%, as measured through Single-Item Self-Rating Adherence Scale (SRSI)
* Own a smartphone

Exclusion Criteria:

* Reside in a nursing home, prison, and/or receiving in-patient psychiatric care at time of enrollment
* Terminal illness with life expectancy <6 months
* Planning to move out of the area in the next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Schnall, PhD, MPH, RN, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Birmingham AIDS Outreach, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Columbia University Irving Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schnall R, Jia H, Brin M, Kay ES, Wood OR, Abua J, Batey DS. Efficacy of CHAMPS for Improving Viral Suppression: A Randomised Clinical Trial. AIDS Behav. 2025 Nov;29(11):3703-3713. doi: 10.1007/s10461-025-04811-x. Epub 2025 Jul 10. PMID 40634827
- [Derived] Wood OR, Schnall R, Kay ES, Jia H, Abua JA, Nichols TK, Olender SA, Mugavero MJ, Batey DS. A community health worker and mobile health app intervention to improve adherence to HIV medication among persons with HIV: the CHAMPS study protocol. BMC Public Health. 2023 May 24;23(1):942. doi: 10.1186/s12889-023-15616-9. PMID 37226141

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 150 | 150
Completed | 113 | 122
Not Completed | 37 | 28
Not completed — Withdrawal by Subject | 11 | 8
Not completed — Lost to Follow-up | 26 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (11.4) | 49.4 (11.9) | 48.1 (11.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 74 | 72 | 146
  Female | 66 | 68 | 134
  Other | 10 | 9 | 19
  Unknown | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic Black | 104 | 115 | 219
  Non-Hispanic White | 17 | 11 | 28
  Hispanic | 22 | 17 | 39
  Non-Hispanic Other | 6 | 4 | 10
  Unknown | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 150 | 150 | 300
Education Level [Count of Participants; unit: Participants]
  Less than high school | 45 | 39 | 84
  High school education/(General Education Development (GED) | 47 | 41 | 88
  Greater than high school | 58 | 69 | 127
  Unknown | 0 | 1 | 1
Sexual Orientation [Count of Participants; unit: Participants]
  Homosexual | 52 | 46 | 98
  Heterosexual | 76 | 77 | 153
  Other | 22 | 23 | 45
  Unknown | 0 | 4 | 4
Viral Suppression [Count of Participants; unit: Participants] — Viral suppression defined as an HIV viral load ≤200 copies/mL
  Participants
    Yes | 104 | 105 | 209
    No | 41 | 37 | 78
    Unknown | 5 | 8 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Virally Suppressed Participants
Description: The number of virally suppressed participants. Viral suppression defined as viral load of <200 copies/mL.
Time Frame: 6 month follow up, 12 month follow up
Population: N=123 intervention (CHAMPS) participants completed the 6 month visit. Of the 123 samples collected, four samples could not be processed by the laboratory, resulting in 119 analyzed. N=113 intervention participants completed the 12 month visit. Of the 113 completers, seven samples could not be processed by the laboratory, resulting in 106 analyzed in the intervention arm. N=116 analyzed in the control arm at month 12, as six samples could not be processed by the laboratory.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 119 | 122
Participants
  6 months | 97 | 94
  12 months: number analyzed (Participants) | 106 | 116
  12 months | 79 | 89

2. Secondary Outcome: Antiretroviral Therapy (ART) Adherence - CleverCap
Description: The CleverCapTM dispenser will automatically record each time a participant opens the dispenser. The investigators will collect adherence data each day from the start to the end of trial (day 1 to 12 months) and report the number of days used.
Time Frame: Up to 12 months
Population: 141 participants analyzed as 141 participants used the CleverCap device and app. Nine participants never used the CleverCap device and app.
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Intervention: Wise App that delivers medication adherence reminders and community health worker sessions Wise App with medication adherence reminders: The Intervention group will receive the Wise App that delivers medication adherence reminders.
  CHW Sessions: The Intervention group will complete sessions with a community health worker (CHW).
Arm/Group | Intervention
Number analyzed (Participants) | 141
Days | 244 (124)

3. Secondary Outcome: Change in Score on the Self-Rating Scale Item (SRSI)
Description: The Self-Rating Scale Item is a single-item self-report adherence measure that uses a 5-point Likert scale to describe medication adherence over the past 4 weeks. Scores range from 1(very poor) to 6 (excellent).
Time Frame: 6 month follow up and 12 month follow up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 113 | 122
score on a scale | 0.04 (0.13) | -0.08 (0.13)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 1/150 | 5/150
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/150
Other Adverse Events (participants affected / at risk) | 0/150 | 0/150

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/49/NCT04562649/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT04562649/ICF_001.pdf